CLINICAL TRIAL: NCT03702452
Title: The Effect and Mechanism of wCST-LL Based Precision Rehabilitation Nursing on Motor Dysfunction After Acute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81871839
Record Dates: First submitted 2018-08-26; First posted 2018-10-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in experimental group were graded with modified Barthel index score, and according to the functional score of patients, the corresponding rehabilitation method was selected for functional rehabilitation from functional rehabilitation nursing program,twice a day with 30 min each time, last 1 week.
  Interventions: Other: functional rehabilitation nursing program
- control group (Experimental): Patients in control group were given conventional bedside rehabilitation ,twice a day with 30 min each time, last 1 week.
  Interventions: Other: control group

INTERVENTIONS:
Other: functional rehabilitation nursing program — According to the modified Barthel index score, the patients' function was divided into four parts Level,each level has different kinds of rehabilitation nursing.
  Arms: Experimental group
Other: control group — The rehabilitation were given by the rehabilitation therapist based on the patient's condition, such as, bridge movement,limb passive motion, limb active motion,turn over,sit upw,walk, and so on.
  Arms: control group

SUMMARY:
Ischemic stroke is the main cause of disability in the world. More than 70% of stroke patients show various degrees of neural function impairment. Motor rehabilitation in acute phase is beneficial for improving patient's structure and function of corticospinal tract. However, it is difficult to obtain effective rehabilitation during the acute phase of stroke because of the insufficiency of professional rehabilitation therapists in stroke wards in China.The present study is to verify that nursing-directed rehabilitation can compensate for the shortage of professional rehabilitation therapists. Our previous study indicated that nursing-directed motor function rehabilitation provided more obvious effect on stroke patients with a weighted corticospinal tract lesion load (wCST-LL) smaller than 2ml. We assume that implementing rehabilitation nursing based on the wCST-LL can realize nursing-directed, wCST-LL-based precision motor rehabilitation during acute phase of ischemic stroke.The present study is to conduct randomized clinical trial to confirm the effect of nursing-directed precision rehabilitation for motor function in acute stroke patients grouped by wCST-LL, and to evaluate the effect of this precision rehabilitation by using functional scale, and to explore the histopathologic mechanism of the precision rehabilitation nursing by mean of neuroelectrophysiology and neuroimaging examination. This study might provide theoretical support for motor rehabilitation in patients during acute phase of stroke.

ELIGIBILITY:
Inclusion Criteria:

* the patients were diagnosed as ischemic stroke by CT or MRI and met the diagnostic criteria of World Health Organization(WHO);
* First stroke, within 7 days, with limb dysfunction (muscle strength < 5 grade);
* there was no contraindication sign of MRI and transcranial magnetic stimulation(TMS) examination, and the examination was completed with good image quality and complete clinical data;
* 18≤ages≤90;
* consciousness

Exclusion Criteria:

* the blood vessels are reconnected after thrombolysis;
* there are serious cardiopulmonary dysfunction, history of craniocerebral trauma, and other diseases affecting the affected side

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of motor function | 0 week and 1 week
  use Modified Barthel scale to evaluate the change of motor function,The scale were measure the function of the stroke patients,the scale have 100 scores,the function is better if the scores were higher.

SECONDARY OUTCOMES:
Change of neuroelectric physiological parameters | 0 week and 1 week
  use the transcranial Magnetic Stimulation to evaluate the function of Corticospinal Tract

OTHER OUTCOMES:
Change of neuroimaging quantitative parameters | 0 week and 12 weeks
  use the Diffusion Weighted Imaging and Diffusion Tensor Imaging to evaluate the function of Corticospinal Tract

CONTACTS AND LOCATIONS:
Overall Officials: jingfen Jin, Master, Principal Investigator — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Chen Y, Zhang Y, Li M, Jin J. Rehabilitation nursing for motor functional recovery of acute ischaemic stroke: study protocol for a randomised controlled trial. BMJ Open. 2020 Sep 25;10(9):e037391. doi: 10.1136/bmjopen-2020-037391. PMID 32978194